CLINICAL TRIAL: NCT05132582
Title: A Randomized, Double-blind, Phase 3 Study of Tucatinib or Placebo in Combination With Trastuzumab and Pertuzumab as Maintenance Therapy for Metastatic HER2+ Breast Cancer (HER2CLIMB-05)
Brief Title: A Study of Tucatinib or Placebo With Trastuzumab and Pertuzumab for Metastatic HER2+ Breast Cancer
Acronym: HER2CLIMB-05
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGNTUC-028; C4251007 (Other: Alias Study Number); 2023-503826-37-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: HER2 Positive Breast Cancer
Keywords: HER2+ breast cancer; Breast Cancer; Metastatic breast cancer; Seattle Genetics
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tucatinib + trastuzumab + pertuzumab (Experimental): Tucatinib + trastuzumab + pertuzumab
  Interventions: Drug: Tucatinib; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Combination product: Trastuzumab + Pertuzumab
- Placebo + trastuzumab + pertuzumab (Active Comparator): Placebo + trastuzumab + pertuzumab
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Combination product: Trastuzumab + Pertuzumab; Drug: Placebo

INTERVENTIONS:
Drug: Tucatinib — 300mg given by mouth (orally) twice daily
  Other Names: TUKYSA, ONT-380, ARRY-380
  Arms: Tucatinib + trastuzumab + pertuzumab
Drug: Trastuzumab — 6mg/kg given into the vein (IV; intravenously) or 600mg injected under the skin (SC; subcutaneous) every 21 days
  Other Names: Herceptin, Herceptin Hylecta
Drug: Pertuzumab — 420mg given by IV every 21 days
  Other Names: Perjeta
Drug: Combination product: Trastuzumab + Pertuzumab — 600 mg pertuzumab, 600 mg trastuzumab, and 20,000 units hyaluronidase will be given by subcutaneous injection every 21 days. May be given in place of trastuzumab and pertuzumab individually.
  Other Names: Phesgo
Drug: Placebo — Given orally twice daily
  Arms: Placebo + trastuzumab + pertuzumab

SUMMARY:
This study is being done to see if tucatinib works better than placebo when given with other drugs to treat participants with HER2-positive breast cancer. A placebo is a pill that looks the same as tucatinib but has no medicine in it. This study will also test what side effects happen when participants take this combination of drugs. A side effect is anything a drug does to the body besides treating your disease.

Participants will have cancer that has spread in the body near where it started (locally advanced) and cannot be removed (unresectable) or has spread through the body (metastatic).

In this study, all participants will get either tucatinib or placebo. Participants will be assigned randomly to a group. This is a blinded study, so patients and their doctors will not know which group a participant is in.

All participants will also get trastuzumab and pertuzumab. These are 2 drugs used to treat this type of cancer.

DETAILED DESCRIPTION:
Control arm: Placebo given orally twice daily plus trastuzumab and pertuzumab every 21 days

Experimental arm: Tucatinib 300 mg given orally twice daily plus trastuzumab and pertuzumab every 21 days

Trastuzumab and pertuzumab will be administered as follows:

• Trastuzumab will be given intravenously (IV) at a dose of 6 mg/kg or subcutaneously (SC) at a fixed dose of 600 mg, once every 21 days.

AND

* Pertuzumab will be given IV at 420 mg every 21 days. OR
* Fixed dose combination of 600 mg pertuzumab, 600 mg trastuzumab, and 20,000 units hyaluronidase will be given SC, once every 21 days, in lieu of trastuzumab and pertuzumab individually.

ELIGIBILITY:
Inclusion Criteria:

* Centrally confirmed HER2+ breast carcinoma according to the 2018 American Society of Clinical Oncologists (ASCO) College of American Pathologists (CAP) guidelines prior to randomization (defined as a 3+ score on immunohistochemistry (IHC) and/or 2+ IHC and concurrent positive by ISH).
* Have unresectable locally advanced or metastatic disease.

  * If recurrent (after [neo]adjuvant therapy), must be at least 6 month treatment free from any trastuzumab and pertuzumab received in the early breast cancer setting for advanced HER2+ disease.
* Have received 4-8 cycles of pre-study induction therapy including only trastuzumab, pertuzumab, and taxane as first-line of therapy for the treatment of advanced breast cancer prior to study enrollment. Participants are eligible provided they are without evidence of disease progression following completion of induction therapy.
* Known hormone receptor status (per local guidelines; may be hormone receptor positive [HR+] or negative [HR-])
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* CNS Inclusion - Based on screening contrast-enhanced brain magnetic resonance imaging (MRI), participants may have any of the following:

  * No evidence of brain metastases
  * Untreated brain metastases which are asymptomatic not needing immediate local treatment and, if identified on prior brain imaging, without evidence of progression since starting first-line induction therapy with trastuzumab, pertuzumab, and taxane
  * Previously treated brain metastases which are asymptomatic

    * Brain metastases previously treated with local therapy must not have progressed since treatment

Exclusion Criteria:

* Prior treatment with any tyrosine kinase inhibitor targeting HER2 and/or epidermal growth factor receptor (EGFR) including pyrotinib, lapatinib, tucatinib, neratinib, and afatinib (except neratinib if given in extended adjuvant setting and ≥ 12 months have elapsed since last neratinib dose prior to start of study drug)
* Unable to undergo contrast-enhanced MRI of the brain
* CNS Exclusion - Based on screening brain MRI and clinical assessment

  * Symptomatic brain metastasis after CNS-directed local therapy
  * Progression of brain metastases since starting first line trastuzumab, pertuzumab, and taxane
  * Ongoing use of systemic corticosteroids at a total daily dose of >2 mg of dexamethasone (or equivalent)
  * Any untreated brain lesion in an anatomic site which may pose risk to participant
  * Known or suspected leptomeningeal disease (LMD)
  * Poorly controlled (>1/week) seizures, or other persistent neurologic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 3 years
  The time from the date of randomization to the investigator assessment of disease progression according to RECIST v1.1 or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  The time from randomization to death from any cause.
PFS by blinded independent central review (BICR) per RECIST v1.1 | Up to approximately 3 years
  The time from the date of randomization to the documented disease progression assessed by BICR according to RECIST v1.1 or death from any cause
Time to deterioration of health-related quality of life (HRQoL) | Up to approximately 3 years
  Will be measured based on patient reported outcomes (PROs) according to the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ C30).
Central nervous system (CNS) PFS | Up to approximately 3 years
  The time from randomization to investigator assessed disease progression in brain (RECIST v1.1), or death from any cause
Incidence of adverse events (AEs) | Through 30 days after last study treatment, approximately 18 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of laboratory abnormalities | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.
Incidence of tucatinib dose alterations | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.
Incidence of trastuzumab dose alterations | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.
Incidence of pertuzumab dose alterations | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.
Maximum concentration (Cmax) | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.
Trough concentration (Ctrough) | Through 30 days after last study treatment, approximately 18 months
  To be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (299):
- United States (73):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Central Arkansas Radiation Therapy Institute Inc d.b.a CARTI, Little Rock, Arkansas
  - UCLA Hematology/Oncology - Beverly Hills, Beverly Hills, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - UCSD Medical Center - Encinitas, Encinitas, California
  - Sulpizio Cardiovascular Center at UC San Diego Health, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UCSD Koman Family Outpatient Pavilion, La Jolla, California
  - UCSD Perlman Medical Offices, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology - Laguna Hills, Laguna Hills, California
  - Administrative Address: UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCSD Medical Center - Bankers Hill, San Diego, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCLA Hematology/Oncology - San Luis Obispo, San Luis Obispo, California
  - UCLA Hematology/Oncology- Santa Barbara, Santa Barbara, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Hematology/Oncology Parkside, Santa Monica, California
  - Clinical And Translational Research Center, Torrance, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Harbor-UCLA Medical Center, Torrance, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - UCSD Medical Center - Vista, Vista, California
  - UCLA Hematology/Oncology- Westlake, Westlake Village, California
  - AdventHealth Altamonte Infusion Center, Altamonte Springs, Florida
  - AdventHealth Medical Group Altamonte(second location), Altamonte Springs, Florida
  - AdventHealth Medical Group Altamonte, Altamonte Springs, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - AdventHealth Medical Group Orlando, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Illinois Hospital and Health Systems (Investigational Drug Pharmacy), Chicago, Illinois
  - University of Illinois Hospital and Health Systems (Outpatient Cancer Center), Chicago, Illinois
  - University of Illinois Hospital and Health Systems, Chicago, Illinois
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Cancer Institute, St Matthews Campus, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Mercy Medical Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Cancer Institute., Kansas City, Missouri
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Grand Island, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Grand Island, Grand Island, Nebraska
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Papillion, Nebraska
  - RWJBarnabas Health- Jersey City Medical Center, Jersey City, New Jersey
  - RWJBarnabas Health- Monmouth Medical Center-Southern Campus, Lakewood, New Jersey
  - RWJBarnabas Health- Cooperman Barnabas Medical Center, Livingston, New Jersey
  - RWJBarnabas Health- Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health-Robert Wood Johnson University Hospital, Somerset, Somerville, New Jersey
  - Steeplechase Cancer Center, Somerville, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey
  - Satellite Infusion Center-Monmouth Medical Center Vantage Point Infusion Center, West Long Branch, New Jersey
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic Cancer Center - Strongsville, Strongsville, Ohio
  - Asplundh Cancer Pavillion, Willow Grove, Pennsylvania
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute- Pharmacy, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University Clinical Trials Unit., Macquarie University, New South Wales
  - Western Sydney Local Health District (WSLHD), Westmead Hospital, Westmead, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - St Andrews Medical Centre, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - St John of God Subiaco Hospital Clinical Trials Unit Bendat Family Comprehensive Cancer Centre, Subiaco, Washington
- Austria (5):
  - Ordination Priv.-Doz. Dr. Michael Hubalek, Schwaz, Other
  - Medizinische Universität Graz, Graz
  - Medizinische Universitat Graz, Graz
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Medizinische Universitat Wien Universitatsklinik Fur Frauenheilkunde, Vienna
- Belgium (4):
  - Jules Bordet lnstituut, Anderlecht
  - Universitair Ziekenhuis Brussel (UZ Brussel), Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique St-Pierre, Ottignies
- Brazil (16):
  - CRIO - Centro Regional lntegrado de Oncologia, Fortaleza, Ceará
  - Hospital Araujo Jorge, Goiânia, Goiás
  - A.C. Camargo Câncer Center, Sao Paulo/SP, Other
  - Hospital Do Cancer De Londrina, Londrina, Paraná
  - Liga Norte-Rio Grandense Contra o Cancer, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa - Hospital do Cancer Mae de Deu, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII, Hospital do Amor de Barretos, Barretos, São Paulo
  - Fundacao Dr Amaral Carvalho, Jaú, São Paulo
  - CEPHO- Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Irmandade da Santa Casa de Misericordia de Porto Alegre centro Multidisciplinar de pesquisa clinica, Porto Alegre/RS
  - Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto
  - ICESP- Instituto do Cancer do Estado de Sao Paulo Octavio Frias de Oliveira, São Paulo
  - Sao Camilo Oncologia, São Paulo
  - Clinica de Pesquisas e Centro de Estudos em Oncologia Ginecologica e Mamária Ltda., São Paulo
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Kelowna, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre integre universitaire de sante et de services sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre Hospitalier de l'Universite de Motreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Chile (5):
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Centro de Investigacion Clínica Bradford Hill, Recoleta, Santiago Metropolitan
  - Clinica Universidad Catolica del Maule, Talca
  - Clinica Alemana Temuco, Temuco
  - James Lind Centro De Investigacion Del Cancer, Temuco
- China (28):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The first Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Medical University (NMU) - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Insitute, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Other
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital Binhai Campus, Tianjin
- Czechia (5):
  - Ustavni lekarna Masarykuv onkologicky ustav, Brno, Other
  - Fakultni Thomayerova nemocnice Onkologicka klinika 1. LF UK a FTN, Praha 4 - Krc, Other
  - Masarykuv Onkologicky Ustav, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole Onkologicka klinika 2. LF UK a FN Motol, Praha 5 - Motol
- Finland (2):
  - Tampere University Hospital, FONK/RSYO, Tampere
  - Tampere University Hospital, Tampere
- France (25):
  - Centre Henri Becquerel / Centre Regional de Lutte Contre le Cancer, Rouen, Brittany Region
  - Institut Bergonie, Bordeaux, Cedex
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-roussillon
  - Institut de Cancerologie de lOuest - Site Rene Gauducheau, Saint-Herblain, Loire-atlantique
  - Institut de Cancerologie de lOuest-Saint Herblain, Saint-Herblain, Loire-atlantique
  - Institut Sainte-Catherine., Avignon, Other
  - Sainte Catherine lnstitut du Cancer Avignon Provence, Avignon, Other
  - Center Georges-Francois Leclerc, Dijon, Other
  - CHU Besancon, Besançon
  - Hopital Avicenne, Bobigny
  - CENTRE FRANCOIS BACLESSE - Service lmagerie medicale, Caen
  - Centre de Lutte contre le Cancer - François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Center Leon Berard, Lyon
  - Institut Regional du Cancer de Montpellier Service lmagerie medicale, Montpellier
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hospices Civils de Lyon, Pierre-Bénite
  - "CARIO - Centre Armoricain de Radiotherapie lmagerie medicate et d'Oncologie -Hopital Prive des, Plérin
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - site St-Cloud, Saint-Cloud
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Institut Curie, Saint-Cloud, Île-de-France Region
- Germany (11):
  - University Hospital Muenster Senology, Münster, North Rhine-Westphalia
  - Universitätsmedizin Mannheim Universitätsfrauenklinik, Manheim, Other
  - Pharmacy:Fortuna Herstellung GmbH, Mannheim, Other
  - "Universitatsklinikum Augsburg Klinik fur Frauenheilkunde und Geburtshilfe", Augsburg
  - Charite Universtitatsmedizin Berlin Klinik fur Gynakologie mit Brustzentrum, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Klinik und Poliklinik fur Frauenheilkunde der Technischen Universitat Munchen, München
  - Universitatsklinikum Ulm Klinik fur Frauenheilkunde und Geburtshilfe, Ulm
  - Universitatsklinikum Wurzburg Frauenklinik und Poliklinik, Würzburg
  - Universitatsklinikum Wurzburg, Comprehensive Cancer Center - Mainfranken (CCCMF), Würzburg
- Greece (5):
  - General Hospital of Athens "Alexandra" Clinical Therapeutics Department, Hematology/Oncology Unit, Athens, Attica
  - University General Hospital of Patras, Oncology Department, Internal Medicine Clinic, Patra, Peloponnese
  - University General Hospital of Larissa, Oncology Clinic, Larissa
  - IASO General Clinic Oncology Clinic, Marousi
  - Metaxa Anticancer Hospital of Piraeus, Pireaus
- Italy (16):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - lstituto Nazionale Tumori IRCCS - Fondazione Pascale U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - IRCCS Ospedale Policlinico, San Martino, Genoa, Liguria
  - ASST Monza Ospedale San Gerardo Centro Ricerca di Fase 1, Monza (MB), Lombardy
  - Humanitas lstituto Clinico Catanese, Catania (CT), Sicily
  - Azienda Ospedaliero Universitaria delle Marche SOD Clinica Oncologica, Torrette, The Marches
  - Divisione Oncologia Medica, Ospedale di Trento - Presidio Ospedaliero (PO) Santa Chiara, Trento, Trentino-Alto Adige
  - SOC Farmacia, Ospedale di Trento - Presidio Ospedaliero (PO), Trento, Trentino-Alto Adige
  - Oncologia Medica Azienda Usl Toscana Nord Ovest - Ospedali Riuniti di Livor, Livorno, Tuscany
  - S.O.C. Oncologia Medica - Nuovo Ospedale di Prato Santo Stefano, Prato, Tuscany
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - SSD Oncologia Medica Addarii - Zamagni, Policlinico Sant'Orsola - Malpighi, Bologna
  - Istituto Clinico Humanitas, Milan
  - Divisione di Senologia Medica; Istituto Europeo di Oncologia, Milan
  - UOC di Oncologia Medica, Azienda Ospedaliero Universitaria (AOU) di Parma, Parma
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia
- Japan (15):
  - Tesshokai Kameda General Hospital, Kamogawa, Chiba
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Naha Nishi Clinic, Naha, Okinawa
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - St. Luke's International Hospital., Chuo-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
- Netherlands (4):
  - Albert Schweitzer Ziekenhuis, Dordrecht, Other
  - Albert Schweitzer Hospital, Doedrecht, South Holland
  - St. Antonius Hospital, Utrecht
  - VieCuri Medsich Centrum, Venlo
- Poland (5):
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Other
  - Narodowy lnstytut Onkologii im. Marii Sklodowskiej-Curie-Panstwowy lnstytut Badawczy, Gliwice, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Salve Medica Apteka Szpitalna, Lodz
  - SP ZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarowskiego w Opolu, Opole
- Portugal (4):
  - Centro Clinico Academico Braga Hospital de Braga, Braga, Other
  - Hospital CUF Descobertas, Lisbon, Other
  - Instituto Portugues de Oncologia de Coimbra Francisco Gentil, EPE (IPO, Coimbra), Coimbra
  - Fundacao Champalimaud, Lisbon
- South Korea (15):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk Nationl University Hospital, Cheongju-si, North Chungcheong
  - Seoul National University Hospital, Seoul, Other
  - Asan Medical Center, Seoul, Other
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Other
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Other
  - Ewha Womans University Mokdong Hospital, Seoul, Other
  - Severance Hospital Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Dong-A University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
- Spain (22):
  - Hospital El Angel Grupo Hla, S.L.U, Málaga, Andalusia
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Virgen De La Arrixaca, EI Palmar, Murcia
  - Fundación Privada Instituto de Investigación Oncológica de Vall Hebron, Barcelona, Other
  - Hospital San Pedro de Alcantara, Cáceres, Other
  - Hospital Universitario Ramon y Cajal, Madrid, Other
  - Hospital Clinico Universitario de Valencia, Valencia, Other
  - Hospital Universitario de Canarias, La Laguna Tenerife, Santa CRUZ DE Tenerife
  - Hospital General Universitario Alicante, Alicante, Valencia
  - Fundacio de Gestio Sanitaria de I'Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundació Hospital Universitari Vall d'Hebron - Institut de Recerca, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Institut Catala d'Oncologia Girona - ICO Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca (Spain Salamanca), Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacion lnstituto Valenciano de Oncologia, Valencia
- Switzerland (3):
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Kantonsspital Baden., Baden
  - Brust-Zentrum AG, Zurich
- Taiwan (13):
  - National Cheng Kung University Hospital, Tainan, Other
  - MacKay Medical Foundation The Presbyterian Church in Taiwan MacKay Memorial Hospital, Taipei, Other
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Other
  - National Taiwan University Hospital, Taipei, R.o.c
  - Chi Mei Medical Center, Tainan, Tainan
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital LinKou, Taoyuan
- United Kingdom (6):
  - Academic Oncology, London, England
  - The Royal Marsden, Sutton, Surrey
  - Finchley Memorial Hospital, London
  - University College London Hospital (UCLH) NHS Foundation Trust, London
  - The Royal Marsden, London
  - Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Dieras V, Curigliano G, Martin M, Lerebours F, Tsurutani J, Savard MF, Jerzak KJ, Hu X, Martins de Aquino Pimentel LC, O'Sullivan CC, Tokunaga E, Okines A, Huang CS, Jacot W, Sohn J, Cronemberger Silva E, Mueller V, Yang S, Granata G, Shen Q, Santarpia L, Hamilton E; HER2CLIMB-05 Investigators. HER2CLIMB-05: A Phase III Study of Tucatinib Versus Placebo in Combination With Trastuzumab and Pertuzumab as First-Line Maintenance Therapy for HER2+ Metastatic Breast Cancer. J Clin Oncol. 2025 Dec 10:JCO2502600. doi: 10.1200/JCO-25-02600. Online ahead of print. PMID 41369677
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTUC-028